CLINICAL TRIAL: NCT00367653
Title: A Phase 3, Randomized, Open-Label, Comparative Trial Of Azithromycin Plus Chloroquine Versus Mefloquine For The Treatment Of Uncomplicated Plasmodium Falciparum Malaria In Africa
Brief Title: Azithromycin Plus Chloroquine Versus Mefloquine In the Treatment of Uncomplicated P. Falciparum Malaria.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A0661155
Record Dates: First submitted 2006-08-21; First posted 2006-08-23 (Estimated); Last update posted 2008-09-16 (Estimated); Status verified 2008-09

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Azithromycin; Chloroquine; Mefloquine

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Azithromycin plus Chloroquine
- 2 (Experimental)
  Interventions: Drug: Mefloquine

INTERVENTIONS:
Drug: Azithromycin plus Chloroquine — Azithromycin 1000 mg by mouth (PO) (two 500 mg tablets) once daily (QD) for 3 days(Days 0, 1, 2) plus chloroquine 600 mg base PO once daily for 3 days (Days 0, 1, 2)
  Other Names: Zithromax
  Arms: 1
Drug: Mefloquine — Mefloquine 1250 mg PO given as a split dose (750 mg [three 250 mg capsules]) initial dose followed by 500 mg PO (two 250 mg capsules) given 6 to 10 hours later on Day 0
  Arms: 2

SUMMARY:
To compare Azithromycin plus Chloroquine versus Mefloquine to treat uncomplicated plasmodium falciparum malaria.

ELIGIBILITY:
Inclusion Criteria:

* Females and males 18 years of age and older with uncomplicated, symptomatic malaria as as indicated by the presence of both of the following:
* Blood smears positive for Plasmodium falciparum asexual parasitemia between 1000 -100,000 parasites
* Documented fever (38.5 C/101.3 F rectal or tympanic; 37.5 C/99.5 F axillary or 38 C/100.4 F oral) or history of fever (as reported by subject) within the prior 24 hours.

Exclusion Criteria:

* Severe or complicated malaria.
* Pregnant or breast-feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2006-11; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The primary objective is to confirm the hypothesis that azithromycin plus chloroquine is noninferior to mefloquine for the treatment of symptomatic, uncomplicated malaria due to P. falciparum in Africa. | duration of trial
The primary endpoint of the study will be the asexual P. falciparum Parasite Clearance Rates (adjusted for molecular testing determining recrudescence, true failures, from reinfection, true cures) at Day 28 in the Parasitologic Per Protocol population. | duration of trial

SECONDARY OUTCOMES:
A secondary objective is to assess the efficacy of azithromycin plus chloroquine. | duration of trial
Additional secondary objectives include an assessment of the safety and tolerability of all treatment regimens. | duration of trial

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- Burkina Faso (2):
  - Pfizer Investigational Site, Ouagadougou, West Africa
  - Pfizer Investigational Site, Nouna
- Pfizer Investigational Site, Navrongo, West Africa, Ghana
- Pfizer Investigational Site, Kisumu, Kisumu County, Kenya
- Mali (2):
  - Pfizer Investigational Site, Bamako, West Africa
  - Pfizer Investigational Site, Bamako
- Pfizer Investigational Site, Senegal, West Africa, Senegal
- Pfizer Investigational Site, Ndola, Zambia

REFERENCES:
- [Derived] Sagara I, Oduro AR, Mulenga M, Dieng Y, Ogutu B, Tiono AB, Mugyenyi P, Sie A, Wasunna M, Kain KC, Djimde AA, Sarkar S, Chandra R, Robbins J, Dunne MW. Efficacy and safety of a combination of azithromycin and chloroquine for the treatment of uncomplicated Plasmodium falciparum malaria in two multi-country randomised clinical trials in African adults. Malar J. 2014 Nov 25;13:458. doi: 10.1186/1475-2875-13-458. PMID 25425434
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661155&StudyName=Azithromycin%20Plus%20Chloroquine%20Versus%20Mefloquine%20In%20the%20Treatment%20of%20%20Uncomplicated%20P.%20falciparum%20Malaria.